CLINICAL TRIAL: NCT02521350
Title: Perioperative Acute Kidney Injury Incidence and Risk Factors in Non-cardiac Surgery
Brief Title: Determination of Perioperative Acute Kidney Injury Incidence
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Acibadem University (Other)
Collaborators: Kadikoy Hospital (Other); Acibadem Atakent University Hospital (Other); Acibadem Fulya Hospital (Other); Acibadem Ankara Hospital (Other); Acibadem Eskişehir Hastanesi (Other); Acibadem Bursa Hospital (Other); Kayseri Acibadem Hospital (Unknown); Acıbadem Adana Hospital (Other); Acibadem Kozyatagi Hospital (Other); Acibadem Kocaeli Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ATADEK 2015-6 /19
Record Dates: First submitted 2015-06-18; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Intensive Care Unit Syndrome
Keywords: Acute Kidney Injury; Surgery; Perioperative care
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Control: - older than 40 years patients with no specific gender, who will stay at least one night in hospital will be included into our study. And cardiovascular, urological surgery patients and patients with known renal insufficiency will be excluded.

SUMMARY:
In the last few years, acute renal injury (AKI) definition has been significantly changed. In the light of the data obtained from multicenter international studies, acute renal injury was redefined according to RIFLE, AKIN and KDIGO criteria. The common criteria of all three criteria in acute renal failure is the increment of level of creatinine as 0.3 mg/dL or 50 % increment of respective basal value of serum creatinine.

In the current study, older than 40 years patients with no specific gender, who will stay at least one night in hospital will be included and cardiovascular and urological surgery patients and patients with known renal insufficiency will be excluded. It was aimed to measure serum creatinine levels in all included patients at baseline and up to 24h after surgery and will be determined acute kidney injury incidence and risk factors according to new criteria.

ELIGIBILITY:
Inclusion Criteria:

* older than 40 years
* no gender specified
* patients who will stay at least one night in hospital
* patient with normal renal function

Exclusion Criteria:

* patient with renal dysfunction and cardiovascular, urological surgery patients

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: older than 40 years, no gender specified, patients who will stay at least one night in hospital except cardiovascular, urological surgery and known renal insufficiency.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in serum creatinine levels at 24h after surgery | Serum creatinine levels will be measured at baseline and up to 24h after surgery
  AKI incidence determination using 50 % or more than 0.3 mg/dL increment of creatinine levels
Correlation with use of drugs before surgery and serum creatinine level at 24h after surgery | Use of drug before surgery and serum creatinine level at 24h after surgery will be correlated.

CONTACTS AND LOCATIONS:
Overall Officials: Fevzi TORAMAN, Prof.Dr., Principal Investigator — Acibadem University

REFERENCES:
- [Result] Susantitaphong P, Cruz DN, Cerda J, Abulfaraj M, Alqahtani F, Koulouridis I, Jaber BL; Acute Kidney Injury Advisory Group of the American Society of Nephrology. World incidence of AKI: a meta-analysis. Clin J Am Soc Nephrol. 2013 Sep;8(9):1482-93. doi: 10.2215/CJN.00710113. Epub 2013 Jun 6. PMID 23744003
- [Result] Ricci Z, Cruz D, Ronco C. The RIFLE criteria and mortality in acute kidney injury: A systematic review. Kidney Int. 2008 Mar;73(5):538-46. doi: 10.1038/sj.ki.5002743. Epub 2007 Dec 26. PMID 18160961